CLINICAL TRIAL: NCT02369991
Title: Treatment of Compound Tibia Fracture With a Microvascular Latissimus Dorsi Flap and the Ilizarov Technique: a Cross-sectional Study of Long-term Outcomes
Brief Title: Treatment of Compound Tibia Fracture With a Microvascular Latissimus Dorsi Flap and the Ilizarov Technique
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jussi Repo, Researcher, Helsinki University Central Hospital
Other Study IDs: 343/13/03/02/2013/4
Record Dates: First submitted 2015-02-18; First posted 2015-02-24 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Reconstructive Surgical Procedure
Keywords: latissimus dorsi flap; bone transport; bone reconstruction; tibia; tibial fracture
MeSH Terms: conditions — Tibial Fractures | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Reconstructive surgery — Patients were treated with free latissimus dorsi flap and bone transport technique

SUMMARY:
This study assesses the long-term results of compound tibial reconstruction treated with a microvascular latissimus dorsi flap and bone transport technique during the last 25 year in Helsinki University central Hospital.

DETAILED DESCRIPTION:
A retrospective review of hospital records was conducted to chart the clinical and operational characteristics of patient. Patients current condition is assessed by applying two function-related (Disabilities of the Arm, Hand and Shoulder, DASH; Lower Extremity Functional Scale, LEFS) and a health-related quality of life (the 15-dimensions, 15D) questionnaires. The patients received the questionnaires by mail. A written informed consent was obtained from the participants. The obtained data was computerized and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age over 15 years.
* Patients with acute compound tibial fracture or sequela treated with free latissimus dorsi flap and bone transport.

Exclusion Criteria:

* Deceased.
* Patients under 15 years of age.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute compound tibial fracture or sequela treated with free latissimus dorsi flap and bone transport
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) | 10-25 years
  Assesses the function of the donor site
The 15-Dimensions Health-Related Quality of Life (HRQoL) instrument. | 10-25 years
  Assesses the HRQoL
Lower Extremity Functional Scale (LEFS) | 10-25 years
  Assesses the function of the reconstructed limb

CONTACTS AND LOCATIONS:
Overall Officials: Erkki J. Tukiainen, PhD, MD, Study Director — Helsinki University Hospital, Department of Plastic and Reconstructive Surgery.
Locations (1):
- Helsinki University Central Hospital, Helsinki, Uusimaa, Finland